CLINICAL TRIAL: NCT01129648
Title: A Randomized, Double-Blind, Multi-center, Placebo-Controlled, Combination Study to Evaluate the Urate-Lowering Activity, Safety, and Potential Pharmacokinetic Interaction of Oral BCX4208 and Allopurinol Administered in Subjects With Gout
Brief Title: Study to Evaluate sUA-Lowering Activity, Safety & PK Interaction of Oral BCX4208 & Allopurinol Admin. in Subjects w/Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX4208-202
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Gout
Keywords: Hyperuricemia, gout
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Allopurinol; ulodesine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- BCX4208 placebo + Allopurinol placebo (Placebo Comparator): Administered daily for 21 days.
  Interventions: Drug: Placebo
- BCX4208 placebo + Allopurinol 100mg (Active Comparator): Administered daily for 21 days.
  Interventions: Drug: Allopurinol
- BCX4208 placebo + Allopurinol 200 mg (Active Comparator): Administered daily for 21 days.
  Interventions: Drug: Allopurinol
- BCX4208 Placebo + Allopurinol 300 mg (Active Comparator): Administered daily for 21 days.
  Interventions: Drug: Allopurinol
- BCX4208 20 mg + Allopurinol Placebo (Experimental): Administered daily for 21 days.
  Interventions: Drug: BCX4208
- BCX4208 20 mg + Allopurinol 100 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 20 mg + Allopurinol 200 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 20 mg + Allopurinol 300 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 40 mg + Allopurinol placebo (Experimental): Administered daily for 21 days.
  Interventions: Drug: BCX4208
- BCX4208 40 mg + Allopurinol 100 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 40 mg + Allopurinol 200 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 40 mg + Allopurinol 300 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 80 mg + Allopurinol Placebo (Experimental): Administered daily for 21 days.
  Interventions: Drug: BCX4208
- BCX4208 80 mg + Allopurinol 100 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 80 mg + Allopurinol 200 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208
- BCX4208 80 mg + Allopurinol 300 mg (Experimental): Administered daily for 21 days.
  Interventions: Drug: Allopurinol; Drug: BCX4208

INTERVENTIONS:
Drug: Placebo — Administered daily for 21 days
  Arms: BCX4208 placebo + Allopurinol placebo
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 placebo + Allopurinol 100mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 placebo + Allopurinol 200 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 Placebo + Allopurinol 300 mg
Drug: BCX4208 — Administered daily for 21 days.
  Arms: BCX4208 20 mg + Allopurinol Placebo
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 20 mg + Allopurinol 100 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 20 mg + Allopurinol 200 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 20 mg + Allopurinol 300 mg
Drug: BCX4208 — Administered daily for 21 days.
  Arms: BCX4208 40 mg + Allopurinol placebo
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 40 mg + Allopurinol 100 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 40 mg + Allopurinol 200 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 40 mg + Allopurinol 300 mg
Drug: BCX4208 — Administered daily for 21 days.
  Arms: BCX4208 80 mg + Allopurinol Placebo
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 80 mg + Allopurinol 100 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 80 mg + Allopurinol 200 mg
Drug: Allopurinol — Administered daily for 21 days.
  Arms: BCX4208 80 mg + Allopurinol 300 mg
Drug: BCX4208 — Adminstered daily for 21 days
  Arms: BCX4208 20 mg + Allopurinol 100 mg; BCX4208 20 mg + Allopurinol 200 mg; BCX4208 20 mg + Allopurinol 300 mg; BCX4208 40 mg + Allopurinol 100 mg; BCX4208 40 mg + Allopurinol 200 mg; BCX4208 40 mg + Allopurinol 300 mg; BCX4208 80 mg + Allopurinol 100 mg; BCX4208 80 mg + Allopurinol 200 mg; BCX4208 80 mg + Allopurinol 300 mg

SUMMARY:
To evaluate safety and efficacy of BCX4208 alone and in combination with allopurinol in subjects with gout.

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, double-blind, multi-center, placebo-controlled study to evaluate efficacy and safety of BCX4208 alone and in combination with allopurinol in approximately 80 subjects with gout. The study is a factorial design, evaluating doses of BCX4208 previously found to be safe and well-tolerated in healthy subjects and subjects with psoriasis and gout. Doses of allopurinol are according to package insert recommendations.

Approximately 80 subjects will be randomized equally to one of 16 treatment groups.

The study will consist of 3 periods: the Screening Period, the Treatment Period, and the Follow-Up Period. The Screening period will be conducted within Day -30 to Day -1, as long as all inclusion and exclusion criteria are satisfied (see Section 8). For subjects receiving urate-lowering therapy; these subjects must discontinue the urate-lowering therapy by Day -14 to assure a washout period of at least 14 days before entering the Treatment Period. Some Screening procedures such as a recording of medical history and clinical laboratory tests performed at Screening only may be performed at any time during the Screening Period (Day -30 to Day -1). Other Screening procedures must be performed within the 7 days prior to the first dose of study drug (i.e., from Day -7 to Day -1); these include: physical examination, height, weight, clinical chemistry (including baseline and qualifying sUA), hematology, and urinalysis evaluations, CD4+, CD8+, CD20+, and CD56+ lymphocyte counts, a serum pregnancy test in females of child-bearing potential, 12-lead ECG, and vital signs assessments. An otherwise qualified subject may have up to 2 repeated determinations of sUA and/or lymphocyte subsets assayed to meet the entry criteria for this study, as long as the qualifying sUA and lymphocyte subsets assays occur 7 or fewer days prior to the first dose of study drug. These assessments will constitute the Baseline assessments for the purpose of comparisons with these same assessments post-dose.

Gout flare prophylaxis with colchicine or naproxen is required to be started prior to the first dose of study drug. Colchicine 0.6 mg once a day will begin at least 7 days prior to Day 1, or naproxen 250 mg twice daily will be started at least 48 hours prior to Day 1. For subjects who discontinue urate-lowering therapy, the required gout flare prophylaxis will begin at or before the cessation of the urate-lowering therapy.

A recording of concomitant medications and AEs will take place from the time of the signing of the Informed Consent Form (ICF) and throughout the duration of the study.

The Treatment Period begins on Day 1. Subjects are to arrive at the study clinic on Day 1 after an overnight fast. After a final review of eligibility criteria, pre-dose vital signs assessments, and BCX4208, allopurinol, and oxypurinol PK blood draw have been performed, subjects will be randomized and administered the first dose of study drug. Subjects will remain in the study clinic for Hour 2, Hour 4, and Hour 8 PK sampling and will return to the study clinic for efficacy and safety evaluations prior to dosing on Days 2, 8, and 15.

Subjects will take study drug daily from Day 1 to Day 21, so that the Day 22 evaluation will occur approximately 24 hours after the last dose of study drug. After the Day 22 evaluation, subjects will enter the Follow-Up Period and will return to the study clinic on Day 29 for safety evaluation. Subjects may resume their prior urate-lowering therapy after the assessments on Day 29.

Subjects who on Day 29 have unresolved treatment-emergent AEs will be followed beyond Day 29 until either resolution of the AE or until clinically stable. This subset of subjects will conclude their study participation at the Day 50 Telephone Safety Follow-Up Contact.

Efficacy will be assessed during the study by means of sUA concentrations. Safety will be assessed during the study by means of physical examination, weight, clinical chemistry, hematology, and urinalysis parameters, absolute CD4+, CD8+, CD20+, and CD56+ lymphocyte counts, 12-lead ECG, vital signs assessments, and AE assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 to <70 years, with screening sUA > 8.0 mg/dL.
2. Diagnosis of gout according to the criteria of the American Rheumatism Association (1977).
3. Be willing and able to take colchicine 0.6 mg per day or naproxen 250 mg twice daily (with proton pump inhibitor if needed) as prophylaxis for gout flares.
4. Be willing to abstain from blood donations from Day -14 to Day 29/Early Termination.
5. Female participants must be sexually abstinent, sterile, post-menopausal, or on stable contraception.

   * Post-menopausal - females greater ≥ 45 years of age whose last menstrual period, including spotting, was > 1 year ago.
   * Stable contraception - now requires a double barrier method, e.g. condom or diaphragm with spermicide.
6. Male participants must be abstinent, vasectomized or using condoms with spermicide with partners meeting female requirements.

Exclusion Criteria:

1. Unable to tolerate allopurinol.
2. Gout Flare during Screening Period that is resolved less than 2 weeks prior to first treatment.
3. Unstable angina, history of symptomatic arrhythmia, or Class III or IV heart failure.
4. ECG Findings: history of congenital long QT syndrome; QTc interval < 350 msec or > 475 msec.
5. Inadequately controlled hypertension (above either or both 150/95 mm Hg).
6. Moderate or severe renal impairment and/or calculated creatinine clearance <60 mL/min (using Cockcroft-Gault formula).
7. ALT or AST > 2.0 x ULN.
8. CD4+ count by flow cytometry (<500 cells/mm3).
9. Hgb <12 g/dL or > 17 g/dL (males) or < 11 g/dL or > 16 g/dL (females).
10. Hct < 37% or > 51% (males) < 33% or > 47% (females).
11. WBC < 3.7 x 109/L or > 11 x 109/L.
12. Positive Pregnancy Test.
13. Females who are pregnant, breastfeeding or planning a pregnancy with the next 4 months.
14. Positive serology for hepatitis B surface antigen or hepatitis C or HIV type I (HIV Ab).
15. Immunocompromised or on systemic immunosuppressant medications (including anakinra) within 14 days of study dosing.
16. Use of azathioprine or 6-mercatopurine within 14 days of study dosing.
17. Use of HCTZ in doses > 50mg per day within 14 days of study dosing.
18. Recipient of any live, attenuated vaccine within 6 weeks of Screening.
19. Receipt of sUA-lowering drugs, ACTH, within 14 days of study dosing.
20. Use of systemic corticosteroids within 4 weeks prior to study dosing.
21. Clinically significant and relevant drug allergies.
22. Chronic or recurrent infections (3 infections at same site) within 12 months.
23. Cancer within 12 months (except nonmelanomatous localized skin cancer.
24. Alcohol or drug abuse.
25. Investigational drug within 30 days of study dosing.
26. Other medical conditions which, in the opinion of the PI, would jeopardize the safety of the study subject or impact the validity of the study results.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To estimate the dose response relationship of BCX4208 when administered as a monotherapy and in combination with allopurinol on sUA. | Day 22

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Scottsdale, Arizona
  - Irvine, California
  - South Miami, Florida
  - Honolulu, Hawaii
  - Boise, Idaho
  - Lexington, Kentucky
  - Frederick, Maryland
  - Olive Branch, Mississippi
  - Billings, Montana
  - Omaha, Nebraska
  - Reno, Nevada
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Duncansville, Pennsylvania
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Dallas, Texas